CLINICAL TRIAL: NCT00974649
Title: Psychosocial Determinants of Continuing or Discontinuing Infertility Treatment: A Psychological Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, Thomas D'Hooghe, Professor, M.D., Phd, University Hospital, Gasthuisberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UZL FWO
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Infertility
Keywords: drop-out; predictors of treatment continuation/discontinuation; IVF/ICSI; infertility; counseling; psychology; Assisted Reproduction; Counselling
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Included in questionnaire study (No Intervention)
  Interventions: Behavioral: self-report questionnaire

INTERVENTIONS:
Behavioral: self-report questionnaire — validated self-report questionnaires on psychosocial determinants

SUMMARY:
The current study aims to explore and analyse the decision making process of couples in regards to continuing or discontinuing infertility treatment. A longitudinal, prospective cohort design is used which allows the monitoring of patients over a longer period of time. Data will be collected quantitatively (questionnaires) as well as qualitatively (in-depth interviews) to allow for a more specific and in depth experience than can be obtained by using a questionnaire study. Innovative aspects of the study include:

1. exploration of determinants of continuing and discontinuing infertility treatment by using a comprehensive psychological theory (both surface and in-depth)
2. exploration of gender differences in the decision making process in continuing or discontinuing treatment
3. longitudinal and prospective arm of the study will allow to gain insight into the 'process'
4. prediction of continuing/discontinuing treatment based on psychological variables.

ELIGIBILITY:
Inclusion Criteria:

* first IVF/ICSI treatment
* sufficient knowledge of Dutch to fill out questionnaires
* heterosexual couples

Exclusion Criteria:

* insufficient knowledge of Dutch
* having had previous IVF/ICSI treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 315 (Actual)
Dates: Start 2007-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
psychological predictors of continuing or discontinuing infertility treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D'Hooghe, M.D., PhD, Study Director — University Hospital Gasthuisberg, Leuven, Belgium; Uschi Van den Broeck, M.A., Principal Investigator — University Hospitals Gasthuisberg, Leuven, Belgium
Locations (1):
- University Hospitals Gasthuisberg, Leuven, Leuven, Belgium

REFERENCES:
- [Result] Van den Broeck U, D'Hooghe T, Enzlin P, Demyttenaere K. Predictors of psychological distress in patients starting IVF treatment: infertility-specific versus general psychological characteristics. Hum Reprod. 2010 Jun;25(6):1471-80. doi: 10.1093/humrep/deq030. Epub 2010 Mar 25. PMID 20338959